CLINICAL TRIAL: NCT05829642
Title: Evaluating the Rollout of Estonia's Enhanced Care Management Program
Brief Title: Estonia's Enhanced Care Management Impact Evaluation
Acronym: ECM
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: World Bank (Other); Georgetown University (Other); Estonia Health Insurance Fund (Unknown)
Responsible Party: Principal Investigator, Kevin Croke, Assistant Professor of Global Health, Harvard School of Public Health (HSPH)
Other Study IDs: P169891
Record Dates: First submitted 2023-02-15; First posted 2023-04-26 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Multi-morbidity; Non-communicable Diseases
Keywords: non-communicable diseases; diabetes; hypertension; obesity; mental health
MeSH Terms: conditions — Noncommunicable Diseases; Diabetes Mellitus; Hypertension; Obesity; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ECM intervention arm: The Enhanced Care Management (ECM) intervention consists of training and coaching family physicians and their teams to develop holistic care and pro-active outreach plans for chronically ill patients or those vulnerable to developing chronically illnesses, as identified and agreed between the enrolled providers and the Estonian Health Insurance Fund (EHIF). The core goal of ECM is to improve the quality of care provided to complex patients, including by increasing the use of preventive care, improving coordination of care across health system levels, and increasing patient involvement in care. These elements can improve patient health and quality of life, and may reduce the need for curative medical services.
  Interventions: Behavioral: Enhanced Care Management
- Control: The control group will not receive any intervention.

INTERVENTIONS:
Behavioral: Enhanced Care Management — ECM aims to enable primary health care providers to coordinate care for patients with complex medical needs. It involves the close coordination of services across all treatment modalities and clinical team members, including primary care physicians, specialists, pharmacists, and other healthcare professionals. Providers undertake:
  Comprehensive care planning: A comprehensive care plan is developed and updated by all members of the patient's healthcare team, including their primary care physician, specialist, and other providers, to ensure that all aspects of treatment are addressed.
  Proactive outreach: Outreach activities, such as phone calls, home visits, and other forms of contact with the patient and their family are also used to promote patient engagement in health management
  Monitoring: Close monitoring of patients and their health conditions is essential to ensure that treatments are effective and that any adverse effects are quickly identified and addressed
  Other Names: ECM coaching
  Groups: ECM intervention arm

SUMMARY:
Estonia's aging population faces an increasing burden of non-communicable diseases (NCDs) and a growing population suffers with multiple chronic conditions. These changes have reduced well-being and quality of life for many older Estonians, while increasing the use of high cost specialist and emergency care. In response, the Estonia Health Insurance Fund (EHIF) is working to support primary care physicians to improve care for complex patients with multiple chronic conditions. A new EHIF-led program, Enhanced Care Management (ECM), entails training family physicians to identify complex patients, co-develop proactive care plans with them, and to undertake more active outreach to and management of these patients.

DETAILED DESCRIPTION:
The Enhanced Care Management (ECM) intervention consists of training and coaching family physicians and their teams to develop holistic care and pro-active outreach plans for chronically ill patients or those vulnerable to developing chronically illnesses, as identified and agreed between the enrolled providers and the Estonian Health Insurance Fund (EHIF). Under ECM, patients covered by EHIF and suffering from chronic diseases such as diabetes and cardiovascular diseases will be proactively engaged and monitored by primary care providers to provide better care and to prevent health deterioration.

Risk-stratified care management for chronic conditions was first introduced in Estonia in 2017 to better support high-risk patients with an assortment of chronic conditions and an increased risk of healthcare utilization. The Enhanced Care Management (ECM) program is intended to improve the quality of care provided to complex patients with qualifying chronic conditions, by increasing the use of preventive care, improving coordination of care across health system levels, and increasing patient involvement in care. These elements can improve patient health and quality of life, and may reduce the need for curative and higher-level medical services-for example, by supporting patients with type 2 diabetes to improve their diet and increase physical activity to limit further deterioration in their health and use of emergency or specialty health services.

In 2017, the World Bank, EHIF and the Estonian Family Physicians Association launched a pilot of risk-stratified care management with a very small number of volunteering primary health care providers. From January to February 2017, a digital environment was developed to monitor patients for family physicians. It contains important data of risk patients (health indicators, medical history, socio-economic background) which can be accessed digitally by health care providers. This allowed family physicians and nurses to monitor health indicators and treatment goals of high-risk patients and track the implementation of the treatment plan.

The family physician and nurse's responsibilities involved assessing patient needs, creating treatment plans, coordinating health-related activities, and working with a social worker to provide social support. During the pilot project, family physicians collaborated with hospitals to track patient outcomes. Results of the initial pilot convinced EHIF that it would be beneficial to test expansion of the ECM model nationally, so a full-scale study was launched during 2020 to include a representative sample of clinics and their eligible patients nationwide.

In this study, the research team will conduct a randomized controlled trial in partnership with EHIF to evaluate the impact of ECM training for physicians. The RCT will have enrolled a randomly selected 97 family physicians out of the 786 family physicians practicing in Estonia. Among those physicians' 6,739 ECM-eligible patients, 2,389 patients will have been randomly selected for enrollment into the ECM program. Using administrative records, the study will evaluate the effects of ECM enrollment on: (1) health care utilization; (2) provider management of tracer conditions; and (3) markers of quality of care such as hospital admission for primary health care-sensitive conditions.

ELIGIBILITY:
Inclusion Criteria:

* identified by general practitioner as having multiple chronic health conditions including type 2 diabetes, hypertension, and obesity

Exclusion Criteria (for patients):

* terminal illness; acute cancer (cancer in treatment), schizophrenia, dialysis due to renal failure, congenital malformations requiring specialized care, and rare diseases; patients with more than 7 chronic conditions

Exclusion Criteria (for clinics) Having participated in ECM pilot study; not being currently operational; or having five or more practicing providers in the clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All clinics and individuals covered by the Estonian Health Insurance Fund and determined to be eligible for Enhanced Care Management
Sampling Method: Probability Sample
Enrollment: 2389 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with primary health care utilization | through study completion, an average of 2 years
  number of primary health care service interactions
Number of Participants with inpatient care interactions | through study completion, an average of 2 years
  number of hospitalizations
Number of Participants with outpatient services | through study completion, an average of 2 years
  number of times ambulatory services accessed
Number of Participants with avoidable hospital admissions | through study completion, an average of 2 years
  number of hospital admissions with asthma, COPD, diabetes, congestive heart failure, or hypertension as primary diagnosis
Number of Participants with emergency department visits | through study completion, an average of 2 years
  number of emergency department visits for any reason
Number of Participants with hospital readmission | through study completion, an average of 2 years
  Inpatient readmission within 90 days after any previous inpatient admission

SECONDARY OUTCOMES:
Number of Participants with inpatient post-hospitalization services | through study completion, an average of 2 years
  number of inpatient post-hospitalization services
Number of Participants with outpatient post-visit services | through study completion, an average of 2 years
  number of outpatient post-visit services
Number of Participants with telephone follow up contacts | through study completion, an average of 2 years
  number of follow up contacts with patient by telephone
Number of Participants with chronic illness-related follow up contacts | through study completion, an average of 2 years
  number of follow up contacts with patient due to chronic illness
Number of diabetes, hypertension and myocardial infarction patients with monitoring of glycosylated Hb (HbA1C) | through study completion, an average of 2 years
  monitoring of glycosylated Hb (HbA1C)
Number of diabetes, hypertension and myocardial infarction patients with monitoring of creatinine | through study completion, an average of 2 years
  monitoring of creatinine
Number of diabetes, hypertension and myocardial infarction patients with monitoring of cholesterol levels and fractions | through study completion, an average of 2 years
  monitoring of cholesterol levels/fractions
Number of hypertension care (high risk patients), diabetes, and myocardial infarction patients | through study completion, an average of 2 years
  counseling
Number of myocardial infarction patients with appropriate statin prescription | through study completion, an average of 2 years
  number of appropriate prescriptions of statins
Number of myocardial infarction patients with appropriate beta-blockers prescription | through study completion, an average of 2 years
  number of appropriate prescriptions of beta-blockers
Number of diabetes patients with appropriate prescriptions | through study completion, an average of 2 years
  number of appropriate diabetes medication prescriptions
Number of participants with hypertension (moderate or high-risk patients) with appropriate drug prescription | from enrollment to study completion
  appropriate drug prescription as defined by EHIF
Number of participants with hyperthyroidism monitoring with TSH adequately measured | through study completion, an average of 2 years
  TSH (thyroid stimulating hormone) determined
Number of participants with new diagnosis of tracer conditions | through study completion, an average of 2 years
  hypertension, Type 2 diabetes, or myocardial infarction diagnosis
Number of participants with prescriptions obtained | through study completion, an average of 2 years
  Share of prescriptions purchased out of all the prescribed medications by provider
Number of participants with inadequate acute care follow up | through study completion, an average of 2 years
  Inadequate follow up care for patients hospitalized for acute inpatient care or surgery: cardiovascular disease, acute myocardial infarction, stroke, hip fracture, cholecystectomy.
Number of participants with incomplete discharge from acute care | through study completion, an average of 2 years
  Incomplete discharge from acute in-patient care (for heart failure, acute myocardial infarction, unstable angina) as defined by EHIF protocol
Number of hypertension patients (all risk levels) with drug prescription appropriate | through study completion, an average of 2 years
  Percentage of active ingredients-based prescriptions

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Croke, Phd, Principal Investigator — Harvard University; Daniel Rogger, PhD, Principal Investigator — World Bank; Benjamin Daniels, MSc, Principal Investigator — Georgetown University
Locations (1):
- Estonia Health Insurance Fund, Tallinn, Harju, Estonia

IPD SHARING:
Plan to Share IPD: Yes
IPD will be anonymized and catalogued on the World Bank Microdata Catalog in consultation with EHIF, including indicators identifying the design variables relevant to each individual.
Supporting Information: Analytic Code
Time Frame: Post-conclusion of analysis; indefinitely.
Access Criteria: Use for research only; per agreement with EHIF.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT05829642/Prot_SAP_000.pdf